CLINICAL TRIAL: NCT04476537
Title: A Phase Ib High-throughput Pancreas Precision Oncology Study Investigating the Feasibility, Efficacy, and Pharmacodynamics of Cell Regulatory-network Analysis Based Therapy Selection in Advanced Pancreatic Adenocarcinoma
Brief Title: RNA Precision Oncology in Advanced Pancreatic Cancer
Acronym: HIPPOCRATES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of feasibility
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Gulam Manji, Associate Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR6703
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic ductal adenocarcinoma (PDA); Precision medicine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention Arm (Experimental): Individuals who meet the eligibility criteria based on their provided tissue sample will be followed by the investigators to obtain medical information every 4 weeks. This follow-up will consist of a review of medical records, contact with the participant's treating physician, or personal contact between the participant and the investigators at Columbia University Irving Medical Center (CUIMC). During the study, their tumor tissue will be evaluated to identify medications that may help treat the cancer. The results of these tests will be reviewed by experts on a Precision Medicine Tumor Board (PMTB) and these experts may recommend a specific treatment to the participant or participant's physician.These participants will continue to be followed until death or withdrawal of consent from the study.
  Interventions: Device: OncoTreat

INTERVENTIONS:
Device: OncoTreat — OncoTreat is a computational pipeline that begins with a tumor expression profile and ends with a list of several candidate regimens.

SUMMARY:
The overall objective of this project is to determinate the feasibility of administering personalized therapy to subjects with advanced pancreatic cancer utilizing the novel OncoTreat platform. The primary objective of this study is to assess the feasibility of implementing the OncoTreat framework in patients with newly diagnosed, untreated metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDA) is a major health problem in the United States and throughout the world. Pancreatic ductal adenocarcinoma (PDA) has the worst prognosis of any major malignancy in the United States and, unlike other common cancers, annual deaths from PDA are rising. During 2017, it is estimated that 53,670 people were diagnosed with PDA and approximately 43,090 people died from PDA in the U.S. Despite recent advances, cytotoxic chemotherapy for PDA has been disappointing with response rates of 20-30% for the most active regimens and little activity for targeted therapies. Even among the small subset of patients who are suitable for surgical resection at the time of diagnosis, complete resection is followed by recurrence in >90% of patients without further systemic therapy, with a median time to recurrence of 6.9 months. Thus all PDA patients require systemic chemotherapy and more effective regimens are urgently needed.

Previous versions of this record contained reference to an observational arm in error. The observational arm has been removed from the record for consistency with the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Age ≥18 years of age on day of signing informed consent.
* Have histologically or cytologically confirmed diagnosis of pancreatic ductal adenocarcinoma or be willing to undergo a biopsy with confirmed pathology prior to starting therapy.
* Have untreated disease that is unresectable due to being metastatic or locally advanced without potential of surgery as assessed by the treating physician.
* Subjects who have documented disease recurrence greater than 6 months after completing neoadjuvant or adjuvant chemotherapy for limited disease will be eligible for the study.
* Have a predicted life expectancy of greater than 6 months.
* Subjects must have a plan to obtain a new core biopsy of a primary and/or metastatic lesion planned as part of routine care for which consent is obtained separately or (b) consent to be biopsied to satisfy the tissue requirements of this protocol.

Exclusion Criteria:

Has previously received neoadjvuant or adjuvant chemotherapy for pancreatic cancer unless greater than 6 months has passed since completion of adjuvant or neoadjuvant chemotherapy and initiation of therapy for recurrent or metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gulam Manji, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen participants enrolled (signed a consent form); however, only one participant started as all others were ineligible or withdrew consent prior to initiation.
Period: Overall Study
Arm/Group | Intervention Arm
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data was not analyzed or disclosed in an effort to protect participant confidentiality (n=1).
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assigned Therapy With OncoTreat
Description: The primary outcome of the study is whether a subject is assigned a therapy that they are able to begin on Part 2 of this study. Assignment of therapy is based on results from OncoTreat analysis and recommendations of the Precision Medicine Tumor Board (PMTB) which included assessment of availability and expected toxicity of identified agents.
Time Frame: 36 months
Population: Data was not analyzed or disclosed in an effort to protect participant confidentiality (n=1).
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 36 months
Description: Data was not analyzed or disclosed in an effort to protect participant confidentiality (n=1).
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT04476537/Prot_SAP_000.pdf